CLINICAL TRIAL: NCT02006056
Title: Prospective Study of Ondissolve in the Prophylaxis/Rescue of Radiation Induced Nausea and Vomiting - a Phase II Study
Brief Title: Ondissolve in the Prophylaxis/Rescue of Radiation Induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Takeda Canada, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Edward Chow, Professor, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ondissolve
Record Dates: First submitted 2013-11-28; First posted 2013-12-09 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Secondary prophylaxis (Experimental): Patients already experiencing mild nausea/vomiting within 24 hours before radiotherapy. Intervention is 8mg of ondansetron (Ondissolve) on the day of radiation treatment at least 1 hour prior to treatment and repeated approx. 608 hours later in the day (bid). For patients who are treated with 20Gy/5 fractions, or 30Gy/10 fractions, they will take ondansetron twice (bid) on each day of treatment, at least 1 hour prior to treatment, and also on weekends or holidays in between treatment.
  Interventions: Drug: Ondansetron
- Primary prophylaxis (Experimental): Patients experiencing no nausea and vomiting 24 hours before commencement of radiotherapy. Intervention is 8mg of ondansetron (Ondissolve) on the day of radiation treatment at least 1 hour prior to treatment and repeated approx. 608 hours later in the day (bid). For patients who are treated with 20Gy/5 fractions, or 30Gy/10 fractions, they will take ondansetron twice (bid) on each day of treatment, at least 1 hour prior to treatment, and also on weekends or holidays in between treatment.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Ondansetron — Patients will take Ondissolve (8mg) on the day of the radiation treatment at least one hour prior to treatment and repeat approximately 6-8 hours later in the day (bid). For patients who are being treated with 20Gy in 5 fractions, or 30 Gy in 10 fractions, this group will take Ondissolve twice (bid) on each day of treatment, at least 1 hour prior to treatment and also on weekends or holidays in between treatment.
  Other Names: Ondissolve

SUMMARY:
The primary objective of the study is to examine the efficacy of Ondissolve for the prevention/rescue of Acute and Delayed Phase radiation induced nausea and vomiting (RINV) in patients undergoing single or multiple fraction, emetogenic palliative radiation therapy for painful bone metastases. The study population will be 30 patients seen in the RRRP at the Sunnybrook Odette Cancer Centre receiving palliative radiation therapy considered emetogenic for bone metastases. Patients will take the study medication (Ondissolve 8 mg) twice on each day of radiation therapy, at least one hour prior to treatment and repeat approximately 6-8 hours later the same day. Patients undergoing multiple fraction radiation therapy will take Ondissolve on weekends or holidays in between treatment. Secondary objectives include to evaluate key secondary endpoints related to RINV, and to investigate the ease and length of administration of protocol medicine. We hypothesize that Ondissolve will be effective in the prophylaxis of RINV, and the ease of use and administration will provide an appropriate delivery method for those unable to tolerate the oral form of ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patient will receive palliative radiation therapy considered emetogenic for bone metastases.
* Group 1: At least mild nausea and/or at least mild vomiting as recorded in the Baseline Nausea and Vomiting Data Collection Sheet
* Group 2: Nausea and vomiting recorded as 'none' in the Baseline Nausea and Vomiting Data Collection Sheet

Exclusion Criteria:

* Patient is scheduled to receive cranial radiation therapy during or within 10 days following completion of protocol RT.
* Patient received cranial RT within 7 days prior to commencement of protocol RT.
* Patient is scheduled to receive chemotherapy during or within 10 days following completion of protocol RT.
* Patient received moderately or highly emetogenic chemotherapy within 7 days prior to commencement of protocol RT.
* Patient is scheduled to change regimen/dose or start the use of corticosteroids (inhaled or topical permitted), or other medications considered to have antiemetic activity within 48 hours of protocol RT.
* Patient is scheduled to change regimen/dose or start the use of corticosteroids (inhaled or topical permitted), or other medications considered to have antiemetic activity during or within 10 days following completion of protocol RT.
* Patient is allergic to protocol medication.
* Patient has a Karnofsky Performance Status score <40.
* Patient is a woman who is pregnant or of childbearing potential and is not using contraceptive measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Chow, MBBS PhD, Principal Investigator — Odette Cancer Centre, Sunnybrook Health Sciences Centre
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients attending the Odette Cancer Centre, Toronto, Canada, who satisfy the eligibility criteria were considered for entry into the trial. The last patient was enrolled July 2014.
Pre-assignment Details: This prospective phase II trial enrolled patients from November 2013 to July 2014.
Groups:
- Primary Prophylaxis: Patients have no pre-existing nausea or vomiting 24 hours before radiotherapy
- Secondary Prophylaxis: Patients already experiencing mild nausea and/or mild vomiting within 24 hours before radiotherapy.
Period: Overall Study
Arm/Group | Primary Prophylaxis | Secondary Prophylaxis
Started | 26 | 4
Completed | 26 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients from both arms received the same treatment, but were divided according to baseline assessment of the presence of nausea or vomiting.
Groups:
- Primary Prophylaxis: Patients had no nausea or vomiting at baseline.
- Secondary Prophylaxis: Patients had nausea or vomiting at baseline.
- Total: Total of all reporting groups
Arm/Group | Primary Prophylaxis | Secondary Prophylaxis | Total
Number analyzed (Participants) | 26 | 4 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.6 (11.7) | 69.8 (5.7) | 71.3 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 1 | 11
  Male | 16 | 3 | 19
Location [Count of Participants; unit: Participants]
  Home | 24 | 4 | 28
  Hospital | 2 | 0 | 2
Score on the KPS [Mean (Standard Deviation); unit: units on a scale] — Karnosky Performance Status Scale: Score from 0-100, with 0 being "dead", and 100 being "Normal no complaints; no evidence of disease"
  units on a scale | 69.2 (15.2) | 70.0 (14.1) | 69.3 (14.8)
Primary cancer site [Count of Participants; unit: Participants]
  Prostate | 10 | 1 | 11
  Breast | 8 | 0 | 8
  Lung | 2 | 1 | 3
  Bladder | 2 | 0 | 2
  Other | 3 | 1 | 4
  Unknown | 1 | 1 | 2
Systemic treatment [Count of Participants; unit: Participants]
  None | 13 | 3 | 16
  Chemotherapy | 7 | 1 | 8
  Hormone therapy | 4 | 0 | 4
  Bisphosphonate only | 2 | 0 | 2
Radiotherapy dose [Count of Participants; unit: Participants]
  8 Gy in 1 fraction | 16 | 4 | 20
  20 Gy in 5 fractions | 6 | 0 | 6
  30 Gy in 10 fractions | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Efficacy for the Prevention/Rescue of Radiation-induced Nausea and Vomiting.
Description: The primary objectives are to examine the efficacy for the prevention/rescue of Acute and Delayed Phase radiation-induced nausea and vomiting (RINV) in patients undergoing single or multiple fraction, emetogenic palliative radiation therapy for painful bone metastases.
  Complete control: No increase in emetic episodes or increase in use of rescue medication (for secondary prophylaxis) following radiation treatment, compared to the number of incidences at baseline.
  Partial control: Increase of 2 or fewer emetic episodes from baseline and no use of rescue antiemetic medication during or after radiotherapy.
  Uncontrolled: Increase of three or more emetic episodes or use of antiemetic rescue medication.
Time Frame: Day 0 - Day 10
Population: The results here encompass the primary outcome measure "the proportion of patients with complete prophylaxis and partial control", which is repeated in the secondary outcome. The secondary outcome "Time to nausea, vomiting and/or use of rescue medication" is unavailable due to the data not being collected/analysed.
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Prophylaxis | Secondary Prophylaxis
Number analyzed (Participants) | 28 | 4
Participants
  Acute-Nausea: number analyzed (Participants) | 26 | 4
  Acute-Nausea: Complete control | 21 | 4
  Acute-Nausea: Partial control | 2 | 0
  Acute-Nausea: Uncontrolled | 3 | 0
  Acute-Vomiting: number analyzed (Participants) | 28 | 2
  Acute-Vomiting: Complete control | 25 | 2
  Acute-Vomiting: Partial control | 1 | 0
  Acute-Vomiting: Uncontrolled | 2 | 0
  Delayed-Nausea: number analyzed (Participants) | 26 | 4
  Delayed-Nausea: Complete control | 18 | 2
  Delayed-Nausea: Partial control | 1 | 0
  Delayed-Nausea: Uncontrolled | 7 | 2
  Delayed-Vomiting: number analyzed (Participants) | 28 | 2
  Delayed-Vomiting: Complete control | 21 | 1
  Delayed-Vomiting: Partial control | 0 | 0
  Delayed-Vomiting: Uncontrolled | 7 | 1
  Combined-Nausea: number analyzed (Participants) | 26 | 4
  Combined-Nausea: Complete control | 17 | 2
  Combined-Nausea: Partial control | 1 | 0
  Combined-Nausea: Uncontrolled | 8 | 2
  Combined-Vomiting: number analyzed (Participants) | 28 | 2
  Combined-Vomiting: Complete control | 21 | 1
  Combined-Vomiting: Partial control | 0 | 0
  Combined-Vomiting: Uncontrolled | 7 | 1

2. Other Pre Specified Outcome: The European Organization for Research and Treatment of Cancer Quality of LIfe Questionnaire - C15 Palliative (C15-PAL), From Day 1-5 of Treatment.
Description: Quality of life as measured by the EORTC QLQ-C15-PAL. For multiple fractions of radiotherapy, the questionnaire will be administered on Day 5 and 10 during treatment when applicable. Since the number of secondary prophylaxis patients was small (n=4), quality of life (QOL) analysis was done with two arms combined. Questions on the C15-PAL were scored on a scale of 0-100, with 0 representing no symptoms but low level of functioning and 100 representing severe symptoms and high degree of functioning.
Time Frame: Day 0-5 during treatment
Population: The primary prophylaxis arm and secondary prophylaxis arm patients were combined and analysed together, because the secondary prophylaxis arm had only 4 patients, which was too low to draw any meaningful conclusions.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- C15-PAL Results: C15-PAL results
Arm/Group | C15-PAL Results
Number analyzed (Participants) | 30
units on a scale
  Pain | 50.6 (31.0)
  Dyspnea | 24.1 (25.0)
  Insomnia | 34.5 (33.9)
  Appetite loss | 36.8 (36.0)
  Constipation | 27.6 (34.6)
  Overall quality of life | 47.7 (24.3)
  Physical functioning | 49.0 (36.2)
  Fatigue | 54.8 (34.4)
  Nausea/vomiting | 5.75 (19.0)
  Emotional functioning | 69.2 (25.8)

3. Other Pre Specified Outcome: The European Organization for Research and Treatment of Cancer Quality of LIfe Questionnaire - C15 Palliative (C15-PAL) on Day 6-10 of Treatment.
Description: as for outcome 2
Time Frame: Day 6-10 of treatment
Population: Combined patients from primary prophylaxis and secondary prophylaxis arms, due to the low number of patients in the secondary prophylaxis arm (n=4).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | C15-PAL Results
Number analyzed (Participants) | 30
units on a scale
  Pain | 49.4 (32.5)
  Dyspnea | 25.9 (31.1)
  Insomnia | 44.4 (33.3)
  Appetite loss | 38.3 (36.6)
  Constipation | 27.1 (34.6)
  Overall quality of life | 47.7 (24.3)
  Physical functioning | 49.0 (36.2)
  Fatigue | 54.8 (34.4)
  Nausea/vomiting | 5.75 (19.0)
  Emotional functioning | 69.2 (25.8)

4. Other Pre Specified Outcome: Functional Living Index-emesis (FLIE) at Day 3, Using Questions 2-9, 11-18 (Q1/Q10 Refer to Nausea/Vomiting and Therefore Are Part of Primary Objectives)
Description: Since the number of secondary prophylaxis patients was small (n=4), quality of life (QOL) analysis was done with two arms combined. Questions on the FLIE are reported from 1-7, with "1" being no symptoms and "not at all" for interference with life, and "7" being "a great deal" of symptom and interference with life.
  Q1-9 are for nausea (N). Q 10-18 are for vomiting (V). All questions refer to "during the past 3 days".
  Q1/10: How much N/V have you had? Q2/11: Has N/V affected your ability to maintain usual recreation or leisure activities? Q3/12: Has N/V affected your ability to make a meal or do minor household repairs? Q4/13: How much has N/V affected your ability to enjoy a meal? Q5/14: How much has N/V affected your ability to enjoy liquid refreshment? Q6/15: How much has N/V affected your willingness to see and spend time with family/friends? Q7/16: Has N/V affected your daily functioning? Q8/17: Degree your N/V imposed hardship on you? Q9/18: Degree on your family?
Time Frame: Day 3
Population: Since the number of secondary prophylaxis patients was small (n=4), quality of life (QOL) analysis was done with two arms combined.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C15-PAL Results
Number analyzed (Participants) | 30
units on a scale
  Q2 nausea affecting leisure activities | 1.31 (0.43)
  Q3 nausea affecting ability to do house work | 1.21 (0.81)
  Q4 nausea affecting enjoyment of meals | 1.40 (1.19)
  Q5 nausea affecting enjoyment of refreshments | 1.17 (0.46)
  Q6 nausea affecting spending time with loved ones | 1.10 (0.40)
  Q7 nausea affecting daily functioning | 1.13 (0.43)
  Q8 nausea imposing personal hardship | 1.20 (0.55)
  Q9 nausea imposing hardship on others | 1.13 (0.51)
  Q11 vomiting affecting leisure activities | 1.03 (0.18)
  Q12 vomiting affecting ability to do house work | 1 (0)
  Q13 vomiting affecting enjoyment of meals | 1.03 (0.18)
  Q14 vomiting affecting enjoyment of refreshments | 1.03 (0.18)
  Q15 vomiting affecting spending time with loved on | 1.03 (0.18)
  Q16 vomiting affecting daily functioning | 1.03 (0.19)
  Q17 vomiting imposing personal hardship | 1.07 (0.25)
  Q18 vomiting imposing hardship on others | 1.03 (0.18)

5. Other Pre Specified Outcome: Functional Living Index-emesis (FLIE) at Day 7, Using Questions 2-9, 11-18 (Q1/Q10 Refer to Nausea/Vomiting and Therefore Are Part of Primary Objectives)
Description: as for outcome 4
Time Frame: Day 7
Population: as for outcome 4
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | C15-PAL Results
Number analyzed (Participants) | 30
units on a scale
  Q2 nausea affecting leisure activities | 1.23 (0.82)
  Q3 nausea affecting ability to do house work | 1.19 (0.69)
  Q4 nausea affecting enjoyment of meals | 1.37 (1.01)
  Q5 nausea affecting enjoyment of refreshments | 1.15 (0.60)
  Q6 nausea affecting spending time with loved ones | 1.19 (0.56)
  Q7 nausea affecting daily functioning | 1.19 (0.56)
  Q8 nausea imposing personal hardship | 1.26 (0.71)
  Q9 nausea imposing hardship on others | 1.22 (0.80)
  Q11 vomiting affecting leisure activities | 1.19 (0.68)
  Q12 vomiting affecting ability to do house work | 1.19 (0.68)
  Q13 vomiting affecting enjoyment of meals | 1.30 (1.2)
  Q14 vomiting affecting enjoyment of refreshments | 1.30 (1.2)
  Q15 vomiting affecting spending time with loved on | 1.15 (0.60)
  Q16 vomiting affecting daily functioning | 1.19 (0.68)
  Q17 vomiting imposing personal hardship | 1.19 (0.56)
  Q18 vomiting imposing hardship on others | 1.12 (0.43)

ADVERSE EVENTS:
Groups:
- Ondissolve: Patients will take Ondissolve (8mg) on the day of the radiation treatment at least one hour prior to treatment and repeat approximately 6-8 hours later in the day (bid). For patients who are being treated with 20Gy in 5 fractions, or 30 Gy in 10 fractions, this group will take Ondissolve twice (bid) on each day of treatment, at least 1 hour prior to treatment and also on weekends or holidays in between treatment.
  Ondissolve: Patients will take Ondissolve (8mg) on the day of the radiation treatment at least one hour prior to treatment and repeat approximately 6-8 hours later in the day (bid). For patients who are being treated with 20Gy in 5 fractions, or 30 Gy in 10 fractions, this group will take Ondissolve twice (bid) on each day of treatment, at least 1 hour prior to treatment and also on weekends or holidays in between treatment.
  Palliative Radiation Therapy: Patient will receive palliative radiation therapy considered emetogenic for bone metastases.
Arm/Group | Ondissolve
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
Small sample size, with most patients having no pre-existing nausea and vomiting. finding need to be confirmed in larger study and perhaps in a randomized trial comparing oral pill formation with ondansetron RDF in the prophylaxis of RINV.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No